CLINICAL TRIAL: NCT03744390
Title: A Single-arm Phase II Multicenter Study of IDH2 (AG-221) Inhibitor in Patients With IDH2 Mutated Myelodysplastic Syndrome
Brief Title: IDH2 (AG 221) Inhibitor in Patients With IDH2 Mutated Myelodysplastic Syndrome
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Groupe Francophone des Myelodysplasies (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GFM-IDEAL Study
Record Dates: First submitted 2018-11-13; First posted 2018-11-16 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Myelodysplastic Syndromes; Leukemia Acute Myeloid
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — enasidenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- AG-221 (Experimental): Subjects enrolled will receive continuous 28-day cycles of AG-221 - 100 mg.
  Interventions: Drug: AG-221

INTERVENTIONS:
Drug: AG-221 — Subjects enrolled will receive continuous 28-day cycles of AG-221 -100 mg.
  Other Names: Enasidenib

SUMMARY:
patients with MDS (Myelodysplastic Syndrome) and mutated IDH2 patients will be treated with AG221 (IDH2 inhibitor)

DETAILED DESCRIPTION:
Myelodysplastic syndrome (MDS) are clonal hematopoietic stem cell disorders characterized by ineffective hematopoiesis leading to blood cytopenia, especially anemia, and often evolving to Acute myeloblastic Leukemia (AML). Main prognostic factors of MDS, for progression to AML and survival, include the number and importance of cytopenias, percent marrow blasts and bone marrow cytogenetic abnormalities. These factors are combined in an International Prognostic Scoring System (IPSS) that distinguishes 4 subgroups with significantly different risk of progression to AML and survival (low, intermediate 1 (int 1), intermediate 2 (int 2), high). Low and int 1 subgroups are often grouped together as "favorable " or low risk MDS, and int 2 and high subgroups are " unfavorable " or high risk MDS.

On the other hand, only 50 to 60% of the patients respond to Azacitidine, and most responders relapse within 12 to 15 months resulting in a median survival of only about 6 months in these patients,. As a result there is a need for new therapies in patients who fail to respond to azacitidine or decitabine and for whom there is currently no establish treatment.

Isocitrate dehydrogenase 1 and 2 (IDH1 and IDH2) are key metabolic enzymes that convert isocitrate to α-ketoglutarate. IDH1/2 mutations define distinct subsets of cancers, including low-grade gliomas and secondary glioblastomas, chondrosarcomas, intrahepatic chol-, and hematologic angiosarcomas c malignancies. Somatic point mutations in IDH1/2 confer a gain-of-function in cancer cells, resulting in the accumulation and secretion in vast excess of an antimetabolite, the D-2-hydroxyglutarate (D-2HG). Overproduction of D-2HG interferes with cellular metabolism and epigenetic regulation, contributing to oncogenesis. Indeed, high levels of D-2HG inhibit alpha-ketoglutarate-dependent dioxygenases, including histone and DNA demethylases, leading to histone and DNA hypermethylation and finally a block in cell differentiation.

preclinical studies have demonstrated that inhibition of IDH1/2-mutant enzymes decreases intracellular D-2-hydroxyglutarate (D-2HG) levels, reverses epigenetic dysregulation, and releases the differentiation block.

AG-221, a selective inhibitor of the IDH2 mutant enzyme Overall, in myeloid malignancies, AG221 have been mainly used in generally heavily pretreated AML, with about 40% of responses in patients with the respective IDH 1 and IDH2 mutations, and a median response duration exceeding 1 year when CR or PR was achieved.

Based on these results, the investigators hypothesize that the IDH2 inhibitor (AG 221) may be an effective therapeutic option in patient with IDH2 mutation-positive myelodysplastic syndrome This is an open-label, single-arm multicenter, phase II study

The efficacy of AG 221 will be studied in 3 different groups of MDS patients with IDH-1 mutation:

* Cohort A:Higher risk MDS (IPSS int-2, high) without response (CR,PR,stable disease with HI) after at least 6 cycles of azacitidine or relapse after a response but without overt progression (defined by at least doubling of marrow blasts, compared to pre azacitidine bone marrow, or by AML progression beyond 30% blasts)
* Cohort B:Untreated higher risk MDS (IPSS int-2, high) without life threatening cytopenias (ie red blood cell (ANC) < 500/mm3 or any recent severe infection and/or platelets below 30,000/mm3 and any bleeding symptom). Azacitidine will be added after 3 cycles of AG-221 in the absence of response
* Cohort C: Lower risk MDS with anemia resistant to erythropoietic stimulating agents (primary or secondary resistance)

ELIGIBILITY:
INCLUSION CRITERIA:

Patients must meet all of the following criteria to participate in the study:

1. Myelodysplastic syndrome according to World Health Organization (WHO) classification including non-proliferative AML up to 29% of Bone marrow (BM) blast
2. Age ≥ 18 years
3. Belonging to one of the following categories:

   1. higher risk MDS (IPSS int-2, high) without response to azacitidine (Complete response (CR),Partial Response (PR), stable disease with HI) after at least 6 cycles , or relapsing after a response but without overt progression (defined by at least doubling of marrow blasts, compared to pre azacitidine bone marrow, or AML progression beyond 30% blasts)
   2. Untreated higher risk MDS (IPSS int-2, high) without life threatening cytopenia including absolute neutrophil count (ANC) <500/mm3 or any recent severe infections and/or platelets below 30,000/mm3 and any bleeding symptom
   3. Lower risk MDS with resistance or loss of response to a previous treatment with epoetin alpha/ beta (≥60000 U/w) or Darbopoetin (≥250 ug/w) given for at least 12 weeks and red blood cell (RBC) transfusion requirement at least 2 U/8 weeks in the previous 16 weeks.
4. Presence of IDH2 mutation in either blood or marrow prior to start of therapy
5. Normal renal function, defined by creatinine less than 1.5 times the upper limit of normal, creatinine clearance (Modification of diet in renal disease) (MDRD) ≥ 50 mL/min.
6. Normal liver function, defined by total bilirubin and transaminases less than 1.5 times the upper limit of normal.
7. Adequate cardiac ejection fraction (>40%)
8. Patient is not known to be refractory to platelet transfusions.Written informed consent.
9. Patient must understand and voluntarily sign consent form.
10. Patient must be able to adhere to the visit schedule as outlined in the study and follow protocol requirements.
11. Eastern Cooperative Oncology Group (ECOG) performance status 0-2 at the time of screening.
12. Female subjects of child-bearing potential must agree to undergo medically supervised pregnancy test prior to starting study drug. The first pregnancy test will be performed at screening (within 7 days prior to first study drug administration), and on the day of the first study drug administration and confirmed negative prior to dosing and Day 1 before dosing all subsequent cycles.
13. Female subjects with reproductive potential must have a negative serum pregnancy test within 7 days prior to the start of therapy. Subjects with reproductive potential are defined as sexually mature women who have not undergone a hysterectomy, bilateral oophorectomy or tubal occlusion or who have not been naturally postmenopausal (i.e., who have not menstruated at all) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months). Females of reproductive potential as well as fertile men and their partners who are female of reproductive potential must agree to abstain from sexual intercourse or to use two highly effective forms of contraception from the time of giving informed consent, during the study and for 120 days (females and males) following the last dose of AG-221. A highly effective form of contraception is defined as hormonal oral contraceptives, injectables, patches, intrauterine devices.

Male patients must :

Agree the need for the use of a condom if engaged in sexual activity with a woman of childbearing potential during the entire period of treatment, even if disruption of treatment and during 3 months after end of treatment.

Agree to learn about the procedures for preservation of sperm before starting treatment

EXCLUSION CRITERIA

A patient meeting any of the following criteria is not eligible to participate in the study:

1. Severe infection or any other uncontrolled severe condition.
2. Significant cardiac disease - New York Heart Association (NYHA) Class III or IV or having suffered a myocardial infarction in the last 6 months.
3. Less than 14 days since prior treatment with growth factors (EPO, G-CSF).
4. Use of investigational agents within 30 days or any anticancer therapy within 2 weeks before the study entry with the exception of hydroxyurea. The patient must have recovered from all acute toxicity from any previous therapy.
5. Subject has a heart-rate corrected QT interval using Fridericia's method (QTcF) ≥ 470 msec or any other factor that increases the risk of QT prolongation or arrhythmic events (e.g., heart failure, hypokalemia, family history of long QT interval syndrome). Subjects with prolonged QTcF interval in the setting of bundle branch block may participate in the study.
6. Active cancer or cancer during the year prior to trial entry other than basal cell carcinoma, or carcinoma in situ of the cervix or breast.
7. Patient already enrolled in another therapeutic trial of an investigational drug.
8. Known HIV infection or active hepatitis B or C.
9. Women who are or could become pregnant or who are currently breastfeeding.
10. Any medical or psychiatric contraindication that would prevent the patient from understanding and signing the informed consent form.
11. Patient eligible for allogeneic stem cell transplantation.
12. Known allergies to AG-221 or any of its excipients.
13. No affiliation to a health insurance system.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2019-04-02 (Actual); Primary Completion 2023-02-18 (Actual); Study Completion 2026-03-18 (Estimated)

PRIMARY OUTCOMES:
Overall hematological response | 6 months
  Overall hematological response

SECONDARY OUTCOMES:
Duration Response | 3 years
  Duration Response
Progression IPSS | 3 years
  Progression IPSS

CONTACTS AND LOCATIONS:
Overall Officials: Lionel ADES, Pr, Principal Investigator — APHP
Locations (22):
- France (22):
  - Hôpital André Mignot, Versailles, LE Chesnay
  - CHU Montpellier St Eloi, Montpellier, Montpellier
  - CH d'Angers/Service des Maladies du sang, Angers
  - centre hospitalier Victor Dupouy, Argenteuil
  - CH de la Cote Basque, Bayonne
  - CHU de Bordeaux, Bordeaux
  - CHU Côte de Nacre/Service d'Hématologie Clinique, Caen
  - Hôpital Henri Mondor, Créteil
  - CHU de Grenoble, Grenoble
  - CH Le Mans/Service d'hématologie Oncologie, Le Mans
  - CH lyon, Lyon
  - Institut Paoli Calmettes/Unité d'Hématologie 3, Marseille
  - GHR Mulhouse Sud-Alsace, Mulhouse
  - CHU Nantes - Hôtel Dieu/Service d'Hématologie Clinique, Nantes
  - Hôpital Archet 1/Service d'Hématologie Clinique, Nice
  - CHU de Nimes, Nîmes
  - Hôpital Saint Louis - Service d'hématologie séniors, Paris
  - Hôpital saint Antoine, Paris
  - Centre Henri Becquerel/Département d'Hématologie, Rouen
  - Institut de cancérologie Lucien Neuwirth Saint priest en Jarez, Saint-Priest-en-Jarez
  - Médecine Interne/IUCT Oncopole, Toulouse
  - CHU de Tours, Tours

IPD SHARING:
Plan to Share IPD: No